CLINICAL TRIAL: NCT02812082
Title: Developing and Assessing the Feasibility of Implementing a Video Web-based Patient Education Application
Brief Title: Web-based Patient Education Program to Manage Side Effects of Allogeneic Stem Cell Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is leaving MSK.
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-769
Record Dates: First submitted 2016-06-20; First posted 2016-06-23 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Allo-SCT Patients; Adult Allo-SCT Survivor
Keywords: Web-based; patient education application; 16-769
MeSH Terms: interventions — Surveys and Questionnaires

ARMS (1):
- video web-based patient education application (Experimental): This is a single-arm design. Development of the web-based application will occur over a 6 month period. Patient accrual will not occur until development of the program is complete. Controlled usability testing during the development/design process of the computer program will not be employed as we do not aim to assess the mechanics of patient use, but rather overall time spent interacting with the application in an uncontrolled environment. Following completion of the tool, patient accrual will occur over a six month time period in order to meet our target sample size of up to 50 participants. Participants will be directed to complete a pre-test questionnaire at the time of accrual and will have 3 months to use the program before being directed to complete the post-test questionnaire.
  Interventions: Other: web-based patient education; Behavioral: questionnaire

INTERVENTIONS:
Other: web-based patient education
Behavioral: questionnaire

SUMMARY:
The purpose of this study is to develop an interactive web-based patient education program to help educate patients about the increased risk of MS and its cardiac risk factors following allo-SCT and to inform and motivate patients how to make lifestyle changes. This program will be used in addition to counseling at participants clinic visits. The investigators are not changing the recommendations for prevention and management of these conditions, but rather are trying to improve the way they provide this education to patients.

ELIGIBILITY:
Inclusion Criteria:

* The option to participate will be offered to male and female allo-SCT patients at MSK ≥ 21 years of age who are greater than 90 days post-transplant and followed in or referred to the adult allo-SCT survivorship clinic at MSK
* The option to participate will be offered to male and female allo-SCT patients at MSK ≥ 21 years of age who are greater than 90 days post-transplant and disease free, but have not yet been referred to the survivorship clinic
* Able to understand written and oral English

Exclusion Criteria:

* Patients less than 90 days post-transplant
* Patients without internet access
* Adult post-transplant patients who have relapsed prior to study recruitment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients that use the application | 1 year
  A successful trial will be when ≥ 50% of enrolled patients use the application.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Mosesso, NP, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/